CLINICAL TRIAL: NCT01697514
Title: A Phase 1 Trial of LY2940680 in Pediatric Patients With Recurrent or Refractory Rhabdomyosarcoma or Medulloblastoma
Brief Title: A Study of LY2940680 in Pediatric Medulloblastoma or Rhabdomyosarcoma
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Trial stopped early for poor accrual.
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14492; I4J-MC-HHBD (Other: Eli Lilly and Company)
Record Dates: First submitted 2012-09-28; First posted 2012-10-02 (Estimated); Last update posted 2013-08-27 (Estimated); Status verified 2013-08

CONDITIONS: Medulloblastoma, Childhood; Rhabdomyosarcoma
Keywords: recurrent medulloblastoma
MeSH Terms: conditions — Medulloblastoma; Rhabdomyosarcoma | interventions — LY2940680

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part A: LY2940680 (Dose Escalation) (Experimental): LY2940680 administered orally once daily at escalating doses (92.5 milligrams per square meter [mg/m^2] up to 370 mg/m^2) for two 28 day cycles. Lower dose levels (23 mg/m^2 and 46 mg/m^2) may also be explored, if necessary. Participants receiving benefit may continue until disease progression, unacceptable toxicity, or discontinuation.
  Interventions: Drug: LY2940680
- Part B: LY2940680 (Dose Confirmation) (Experimental): LY2940680 administered orally once daily for two 28 day cycles. Dose based on Part A. Participants receiving benefit may continue until disease progression, unacceptable toxicity, or discontinuation.
  Interventions: Drug: LY2940680

INTERVENTIONS:
Drug: LY2940680 — Capsule administered orally.
Drug: LY2940680 — Powder administered orally (may be sprinkled on soft food).

SUMMARY:
The purpose of this study is to find a recommended dose level of LY2940680 that can be safely given to children with medulloblastoma or rhabdomyosarcoma that has returned or doesn't respond to initial treatment. The study will also explore the changes in a cancer marker levels. Finally, the study will help document any antitumor activity.

ELIGIBILITY:
Inclusion Criteria:

* For Part A: Have a diagnosis of recurrent or refractory rhabdomyosarcoma or medulloblastoma and have had histologic verification of malignancy at original diagnosis or relapse.
* For Part B: Have a diagnosis of recurrent or refractory medulloblastoma and have had histologic verification of malignancy at original diagnosis or relapse.
* Current disease state must be one for which there is no known curative therapy or therapy proven to prolong survival with an acceptable quality of life.
* Karnofsky score must be at least 50% for participants >16 years of age, and Lansky score must be at least 50% for participants 16 years of age or less. Participants who are unable to walk because of paralysis, but who are in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.
* Have fully recovered from the acute toxic effects of all prior anticancer chemotherapy.

  * Participants with solid tumors must not have received myelosuppressive chemotherapy within 3 weeks of enrollment in this study (6 weeks, if previously treated with nitrosourea).
  * Hematopoietic growth factors: At least 14 days after the last dose of a longacting growth factor (eg, Neulasta®) or 7 days for short-acting growth factor.
  * Biologic (antineoplastic agent): At least 7 days after the last dose of a biologic agent.
  * Immunotherapy: At least 6 weeks since the completion of any type of immunotherapy (eg, tumor vaccines).
  * Monoclonal antibodies: At least 3 half-lives of the antibody after the last dose of a monoclonal antibody.
  * Radiation therapy (XRT): ≥8 weeks for local irradiation to primary tumor;≥2 weeks prior to study entry for focal irradiation for symptomatic metastatic sites; ≥3 months for craniospinal XRT, or ≥24 weeks if ≥50% radiation of pelvis; minimum of 6 weeks must have elapsed if other substantial bone marrow radiation has been received.
  * Stem cell transplant: allowed if they have recovered from all acute toxicity and adequate bone marrow reserve is demonstrated. At least 8 weeks must have elapsed since autologous stem cell transplantation or ≥3 months for allogenic transplantation. Participants must be off all immunosuppressive therapy and have no evidence of active graft-versus-host disease.
* Have adequate organ function, including:

  * Bone marrow: Peripheral absolute neutrophil count (ANC) ≥500/cubic millimeter (mm^3) and platelet count ≥100,000/mm^3 (transfusion independent, defined as not receiving platelet transfusions within a 7-day period prior to enrollment).
  * Hepatic: Bilirubin (sum of conjugated + unconjugated)≤1.5 × upper limit of normal (ULN) for age. Serum alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.0 times ULN for age. Serum albumin ≥2 grams/deciliter (g/dL).
  * Renal: Creatinine clearance or radioisotope glomerular filtration rate (GFR)

    ≥70 milliliters/minute/1.73 square meters (mL/min/1.73 m^2), or a serum creatinine based on age/gender per the Schwartz formula for estimating GFR utilizing child length and stature data published by the Centers for Disease Control and Prevention (CDC).
  * Neurologic: Participants with seizure disorders may be enrolled if receiving nonenzyme-inducing anticonvulsants and if the symptoms are well controlled. They must have a stable neurologic status for at least 1 week prior to enrollment in the study.
* Must be able to swallow powder or a capsule.
* Have the presence of either measurable or nonmeasurable disease.

Exclusion Criteria:

* Have received treatment within 21 days of the initial dose of study drug with an experimental agent for noncancer indications that has not received regulatory approval for any indication.
* Receiving corticosteroids and have not been on a stable or decreasing dose of corticosteroid for the prior 7 days.
* Receiving enzyme-inducing anticonvulsants.
* Have serious preexisting medical conditions.
* Have current hematologic malignancies or acute or chronic leukemia.
* Have a known active fungal, bacterial, and/or known viral infection, including human immunodeficiency virus (HIV) or viral (A, B, or C) hepatitis (screening is not required).
* Have a second primary malignancy that, in the judgment of the investigator and sponsor, may affect the interpretation of results.
* Have ≥Grade 2 QT prolongation, that is, QTc interval of >480 milliseconds (msec) on screening electrocardiography (ECG).

Ages: 12 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2013-07; Primary Completion 2016-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose of LY2940680 | Baseline to Part A Completion (estimated as 12 months)

SECONDARY OUTCOMES:
Pharmacokinetics: Area Under the Concentration - Time Curve (AUC) of LY2940680 and LSN2941091 | Predose up to 24 hours Postdose
Pharmacokinetics: Maximum Concentration (Cmax) of LY2940680 and LSN2941091 | Predose up to 24 hours Postdose
Pharmacokinetics: Time of Maximal Concentration (Tmax) of LY2940680 and LSN2941091 | Predose up to 24 hours Postdose
Number of Participants with Tumor Response | Baseline to Study Completion (estimated as 44 months)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (4):
- United States (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Diego, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aurora, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cincinnati, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Portland, Oregon